CLINICAL TRIAL: NCT01500759
Title: Prevalence, Clinical Characteristics and Type of Sleep-disordered Breathing in Patients With Chronic, Symptomatic, Systolic Heart Failure
Brief Title: Sleep-Disordered Breathing in Heart Failure - The SchlaHF-Registry
Acronym: SchlaHF
Status: Completed | Type: Observational
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Other Study IDs: 001
Record Dates: First submitted 2011-12-23; First posted 2011-12-28 (Estimated); Results first posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-05

CONDITIONS: Congestive Heart Failure; Left Ventricular Systolic Dysfunction
Keywords: chronic heart failure; heart failure; hf; sleep-disordered breathing; sdb; nyha; lvef; cheyne stokes; central sleep apnoea; sleep apnoea
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left; Sleep Apnea Syndromes; Cheyne-Stokes Respiration; Sleep Apnea, Central

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective target of the registry is to investigate the prevalence of SDB as well as the clinical characteristics of patients with and without SDB as well as the predominant type of sdb.

For this purpose data from patients suffering from chronic, symptomatic heart failure with impaired left ventricular ejection fraction will be collected prospectively.

DETAILED DESCRIPTION:
Despite recent advances in pharmacological treatment, congestive heart failure (CHF) continues to cause debilitating symptoms, frequent hospital admissions and a high mortality. Despite of therapy with beta-blockers and ACE-inhibitors many patients have persistent symptoms and most will eventually die of cardiovascular causes, often from progressive heart failure.

Sleep Disordered Breathing (SDB) is known to cause consequences, which have negative effects on heart failure.

Objective target of the registry is to investigate the prevalence of SDB, clinical characteristics, symptoms and the degree and type of SDB in patients with chronic HF.

For this purpose data from patients with chronic heart failure will be collected prospectively.In the registry several cardiologists in private practice or hospital and cooperating sleep laboratories shall participate.

Cardiologists screen patients with Chronic Heart Failure (chronic HF) prospectively. In case of suffering from chronic HF for at least 12 weeks since diagnosis, with NYHA III-IV or NYHA class II with at least one hospitalisation for HF in the last 12 months. Written informed consent for data privacy aspects must be obtained before screening for SDB. Patients who satisfy to all inclusion- and exclusion criteria will be included consecutively into the registry.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be over 18
* Chronic heart failure (at least 12 weeks since diagnosis) according to the current applicable guidelines
* Left ventricular systolic dysfunction (LVEF ≤ 45% by imaging method such as echocardiography, radionuclide angiography, left ventriculography, or cardiac magnetic resonance imaging) documented less than 12 weeks
* NYHA class III or IV at the time of inclusion or NYHA class II with at least one hospitalisation for HF in the last 24 months
* Patient is able to fully understand study information and signed informed consent

Exclusion Criteria:

* Life expectancy < 1 year for diseases unrelated to chronic HF
* Cardiac surgery, Percutaneous coronary intervention (PCI), Myocardial Infarction (MI) or unstable angina within 6 months
* CRT-implantation (either CRT-D or CRT-P) scheduled or within 6 months
* Transient ischemic attack (TIA) or Stroke within 3 months
* Hemodynamically significant uncorrected primary valvular heart disease, obstructive or regurgitant, or any valvular disease expected to lead to surgery
* Acute myocarditis/pericarditis within 6 months
* Current CPAP or bilevel therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with Chronic Heart Failure with LVEF ≤ 45% and NYHA III-IV or NYHA class II with at least one hospitalisation for HF in the last 24 months.
Sampling Method: Probability Sample
Enrollment: 6876 (Actual)
Dates: Start 2007-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erland Erdmann, Prof, Principal Investigator — Klinikum der Universität zu Köln; Helmut Teschler, Prof, Principal Investigator — Ruhrlandklinik Essen; Holger Woehrle, MD, Study Director — ResMed
Locations (199):
- Australia (7):
  - Westmead Hospital, Westmead, New South Wales
  - Rivercity Private Hospital, Auchenflower, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Baker IDI Heart and Diabetes Institute, Melbourne, Victoria
  - St Vincents and Mercy Private Hospital, Melbourne, Victoria
  - Melbourne Sleep Disorders Centre, East Melbourne, Victoria 3002
  - Hollywood Private Hospital (CVS), Nedlands, Western Australia
- Germany (192):
  - Cardiopraxis Ingelheim, Ingelheim, Rhineland-Palatinate
  - Praxis Dr. Frieske, Aachen
  - Universitätsklinikum Aachen, Aachen
  - DRK Krankenhaus, Alzey
  - Gemeinschaftspraxis Weiß/ Dr. Heesing, Arnsberg
  - Zentralklinikum Bad Berka, Bad Berka
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Klinik Lazariterhof, Bad Krozingen
  - Praxis Dr. Bauer, Bad Mergentheim
  - HDZ NRW, Bad Oeynhausen
  - Kardiologische Praxis Dr. Stroh, Bad Wurzach
  - Oberlausitz-Kliniken gGmbH, Bautzen
  - Kardiopraxis Rheinberg, Bergisch Gladbach
  - Charité Campus Mitte CCM, Berlin
  - Charité Campus Mitte, Berlin
  - Praxis Gemeinschaft Frille, Berlin
  - POLIKUM Friedenau, Berlin
  - Gemeinschaftspraxis Groß-Ziethener Chaussee, Berlin
  - Unfallkrankenhaus Berlin, Berlin
  - Jüdisches Krankenhaus Berlin, Berlin
  - Charité Campus Virchow Klinikum, Berlin
  - Charité Campus Virchow-Klinikum, Berlin
  - Praxis Westend, Berlin
  - Herzzentrum Brandenburg, Bernau
  - Praxis für Lunge,Herz und Schlaf, Bielefeld
  - Kardiologie Gemeinschaftspraxis Dr. Tenholt, Bochum
  - Universitätsklinikum Bergmannsheil, Bochum
  - Augusta Krankenanstalten Bochum, Bochum
  - St.-Josephs-Hospital, Bochum
  - Kardiologie Kemnade, Bochum
  - Kardiologische Praxis Dr. Staubach, Bochum
  - Praxis für Kardiologie Bonn, Bonn
  - Universitätsklinikum Bonn, Bonn
  - Kardiologische Praxis Marschner, Bonn
  - Gemeinschaftspraxis Kardiologie, Bottrop
  - Gemeinschaftspraxis Dres. Tinnefeld, Bottrop
  - Kardiologie Bühl, Brühl
  - Mediclin Rehazentrum Spreewald, Burg
  - Gemeinschaftspraxis Kardiologie Dr. Becker, Castrop-Rauxel
  - Kardiologische Praxis Dr. Isbruch, Castrop-Rauxel
  - MVZ am Küchwald, Chemnitz
  - Klinikum Coburg GmbH, Coburg
  - St.-Vinzenz Hospital, Cologne
  - Kardiologische Praxis Dr. Fritsch, Cologne
  - Malteser Krankenhaus St. Hildegardis, Cologne
  - Klinikum der Universität zu Köln- Herzzentrum, Cologne
  - Prof. Franzen Institut, Cologne
  - Universitätsklinikum Köln-Herzzentrum, Cologne
  - Praxis Dr. Anselm Bäumer, Cologne
  - Gemeinschaftspraxis Dres. Gysan/Heinzler/May, Cologne
  - Fachkrankenhaus Coswig, Coswig
  - Carl-Thiem-Klinikum gGmbH, Cottbus
  - Praxis Dr. Hecker, Dortmund
  - Kardiologie - Gemeinschaftspraxis Dortmund, Dortmund
  - Kardiologie-Gemeinschaftspraxis Dortmund, Dortmund
  - Kardiologische Praxis Dr. Golling, Dortmund
  - Klinikum Dortmund gGmbH, Dortmund
  - Clinical Trial Site Services, Dortmund
  - Kardiologische Praxis Dr. Wetzel, Dortmund
  - Kardiologische Praxis Dr. Lodde, Dortmund
  - Kardiologische Praxis Dr. Dröse, Dortmund
  - Facharztzentrum Dresden-Neustadt GbR, Dresden
  - Gemeinschaftpraxis Dres. Schmidt/Gronke, Dresden
  - Praxis Dr. Hohensee, Dresden
  - Herzzentrum Universität Dresden, Dresden
  - goMedus Gesundheitszentrum, Düsseldorf
  - Kardiologische Praxis Dr. Horowitz, Düsseldorf
  - Kardiologische Praxis Dr. Raff, Düsseldorf
  - Florence-Nightingale Krankenhaus, Düsseldorf
  - Khs Florence-Nightingale, Düsseldorf
  - Kardiologie Oberkassel, Düsseldorf
  - Gemeinschaftspraxis PD Dr. Lankisch, Düsseldorf
  - Fachärzte für Innere Medizin Dres Ritter, Richter, Mehrer, Kahl, Emmendingen
  - Helios Klinikum Erfurt-Kardiologie, Erfurt
  - Helios Klinikum Erfurt-Schlafmedizin, Erfurt
  - Universitätsklinikum Erlangen, Erlangen
  - Westdeutsches Herzzentrum, Universitätsklinikum Essen, Essen
  - Kardiologische Praxis Dr. Cord Müller, Essen
  - Schwerpunktpraxis Kardiologie Drs. Ophoff/Fritzsch, Essen
  - Kardiologische Praxis Prof. Winter, Essen
  - Kardiologie Praxis Dr. Bonnekamp, Essen
  - Praxis Dr. Tekiyeh, Essen
  - Elisabeth-Krankenhaus Essen, Essen
  - Ruhrlandklinik Essen, Essen
  - Praxis Dr. Rau, Essen
  - Kath. Kliniken Essen / Philippusstift, Essen
  - Gemeinschaftspraxis Dres. Guckenbiehl, Flonheim
  - Kardiologische Praxis Dr. Kruse, Forst
  - CardioVasculäres Centrum Frankfurt, Frankfurt
  - Praxis Dr. Diedrichs, Frechen
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Gemeinschaftspraxis Dres. Böhmeke/Schmidt, Gladbeck
  - Kardiologische Praxis Dr. Hug, Günzburg
  - Kardiologische Praxis Gütersloh, Gütersloh
  - Gemeinschaftspraxis Dres Leischik/Littwitz, Hagen
  - Kardiologische Praxis Dr. Arens, Hagen
  - Gemeinschaftspraxis Dres. Subin/Lutter, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik Barmbek, Hamburg
  - Internistenpraxis Alstertal Hamburg, Hamburg
  - Kardiologische Praxis Dr. Schröder, Hamburg
  - Kardiologische Praxis Dr. Cierpka, Hanover
  - Praxis Dr. Hötte, Hanover
  - Siloah Krankenhaus, Hanover
  - Kardiologische Praxis Dr. Hartung, Hanover
  - Heidelberger Praxisklinik für Kardiologie, Heidelberg
  - Praxis Dr. Durak, Heidelberg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - Evangelisches Krankenhaus Herne, Herne
  - EvK Herne, Herne
  - Kardiologische Praxis Dr. Furche, Herne
  - Gemeinschaftspraxis Dr. Bruch, Herne
  - Kardiologische Praxis Dr. Schlichting, Herne
  - St. Elisabeth-Hospital Herten gGmbH, Herten
  - Praxis für Innere Medizin/Kardiologie, Hoyerswerda
  - Gemeinschaftspraxis Dres. Dobler/Turin, Karlstadt am Main
  - Ambulantes Herzzentrum Kassel, Kassel
  - Kardiologische Praxis Dr. Siegfried Frickel, Kempen
  - Klinik Kitzinger Land, Kitzingen
  - Klinikum Dahme-Spreewald GmbH, Königs Wusterhausen
  - Praxis Dr. Krater, Krefeld
  - Helios Klinikum Krefeld, Krefeld
  - Universitätsklinikum Leipzig-Herzzentrum, Leipzig
  - Helios Krankenhaus Leisnig, Leisnig
  - Gemeinschaftspraxis Dr. Hilgedieck/Sava, Lengerich
  - Kardiologische Praxis Dr. Faber, Lindlar
  - Ärztezentrum Holthausen-Biene, Lingen
  - Kardiologische Praxis Ludwigsburg, Ludwigsburg
  - Universitätsklinikum Schleswig-Holstein Campus Lübeck-Kardiologie, Lübeck
  - Klinikum der Johannes Gutenberg-Universität Mainz, Mainz
  - Gemeinschaftspraxis Dres. Heifer/Loster/Schernus, Mannheim
  - Gemeinschaftspraxis für Herz & Gefäße, Mannheim
  - Universitätsklinik Mannheim-Kardiologie, Mannheim
  - Gemeinschaftspraxis Dres. Brandt / Jakobs, Mannheim
  - Universitätsklinikum Gießen/Marburg Standort Marburg-Kardiologie, Marburg
  - Praxis Dr. Schnabel, Meissen
  - Gemeinschaftspraxis Dr. Jocham, Memmingen
  - Praxis für Kardiologie Dr. med. Menz, Menden
  - Herz-& Gefäßpraxis, Metzingen
  - Praxis Kutenhausen, Minden
  - Krankenhaus Bethanien, Moers
  - Kardiologische Praxis Dr. Schön, Mühldorf
  - Evangelisches Krankenhaus Mülheim, Mülheim
  - Kardiologie am Rotkreuzplatz, München
  - Gemeinschaftspraxis Dres. Wauer / Windstetter, München
  - Kardiologische Praxis Dr. Herholz, München
  - Klinikum Augustinum München, München
  - Praxis Dres. Böhme/Linke, München
  - Kardiologische Praxis Dr. Muradi, Münster
  - Universitätsklinikum Münster, Münster
  - Praxis für Kardiologie Dr. med. Hewing, Münster
  - Städtisches Khs Lukas, Neuss
  - Kardiologische Praxis Nienburg, Nienburg
  - Klinikum Nürnberg Süd, Nuremberg
  - Kardiologische Praxis Dr. Gumbrecht, Ochtrup
  - Kardiologische Praxis Dr. Hassler, Plauen
  - Kardiologische Praxis Dr. Wiethölter, Radebeul
  - Praxis für Kardiologie Ratingen, Ratingen
  - Praxis Dr. Fröhlich, Ratingen
  - DRK Krankenhaus Mölln-Ratzeburg, Ratzeburg
  - Ambulantes Cardiovaskuläres Centrum, Ravensburg
  - Gemeinschaftspraxis Dr. Weber/Dr. Feja, Recklinghausen
  - Universitätsklinikum Regensburg, Regensburg
  - Khs St. Adolf Stift, Reinbek
  - Praxis Dr. Hein, Reinbek
  - Kardiologische Praxis Dr. Kleinz, Remscheid
  - Praxis Dr. Nebel, Rheine
  - Praxis Dr. Kestermann, Rheine
  - Kardiologische Praxis Dr. Figura, Rinteln
  - Praxis Dr. Ebeling, Schönefeld
  - Kardiologische Praxis Dr. Heinze, Schwerte
  - Praxisgemeinschaft Cardio-Soest, Soest
  - Facharztzentrum Sonneberg, Sonneberg
  - Kreiskrankenhaus Stollberg GmbH, Stollberg
  - Kardiologische Praxis Dr. Birkenhagen, Stollberg
  - Klinikum Uelzen GmbH, Uelzen
  - Herzklinik Ulm Dr. Haerer und Partner, Ulm
  - Zentrum für Innere Medizin Uni Ulm, Ulm
  - Katharinen Hospital Unna, Unna
  - Kardiologische Praxis Dr. Burkhard-Meier, Viersen
  - Praxis Dr. Gerritsen, Waldkraiburg
  - Fachkliniken Wangen, Wangen
  - Stiftungsklinik Weißenhorn, Weißenhorn
  - Kardiologisch angiologische Gemeinschaftspraxis, Wiesbaden
  - Kardiologische Gemeinschaftspraxis Dr. K. Vorbeck, Wiesbaden
  - Kardiologische Praxis Dr. Vrettos, Witten
  - Kardiologische Praxis Dr. Rudolf/ Dr. Bernhardt, Worms
  - Comprehensive Heart Failure Center, Universitätsklinikum Würzburg, Würzburg
  - Universitätsklinikum Würzburg, Würzburg
  - Evangel. Khs Zweibrücken, Zweibrücken

REFERENCES:
- [Result] Woehrle H, Oldenburg O, Arzt M, Graml A, Erdmann E, Teschler H, Wegscheider K; SCHLA-HF Investigators. Determining the prevalence and predictors of sleep disordered breathing in patients with chronic heart failure: rationale and design of the SCHLA-HF registry. BMC Cardiovasc Disord. 2014 Apr 9;14:46. doi: 10.1186/1471-2261-14-46. PMID 24716484
- [Result] Arzt M, Woehrle H, Oldenburg O, Graml A, Suling A, Erdmann E, Teschler H, Wegscheider K; SchlaHF Investigators. Prevalence and Predictors of Sleep-Disordered Breathing in Patients With Stable Chronic Heart Failure: The SchlaHF Registry. JACC Heart Fail. 2016 Feb;4(2):116-125. doi: 10.1016/j.jchf.2015.09.014. Epub 2015 Dec 9. PMID 26682790
- [Result] Arzt M, Oldenburg O, Graml A, Erdmann E, Teschler H, Wegscheider K, Suling A, Woehrle H; SchlaHF Investigators. Phenotyping of Sleep-Disordered Breathing in Patients With Chronic Heart Failure With Reduced Ejection Fraction-the SchlaHF Registry. J Am Heart Assoc. 2017 Nov 29;6(12):e005899. doi: 10.1161/JAHA.116.005899. PMID 29187390

RESULTS

PARTICIPANT FLOW:
Groups:
- Chronic HF Without SDB: Patients with chronic heart failure (left ventricular ejection fraction ≤45% or New York Heart Association (NYHA) class III or IV or NYHA class II with ≥1 hospitalization within 12 months before inclusion) and no sleep disordered breathing (SDB, Apnoea-Hypopnoea Index AHI ≥15)
- Chronic HF With SDB: Patients with chronic heart failure (left ventricular ejection fraction ≤45% or New York Heart Association (NYHA) class III or IV or NYHA class II with ≥1 hospitalization within 12 months before inclusion) and sleep disordered breathing (SDB, Apnoea-Hypopnoea Index AHI ≥15)
Period: Overall Study
Arm/Group | Chronic HF Without SDB | Chronic HF With SDB
Started | 3686 | 3190
Completed | 3686 | 3190
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronic HF Without SDB | Chronic HF With SDB | Total
Number analyzed (Participants) | 3686 | 3190 | 6876
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (12) | 69 (11) | 67 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 932 | 516 | 1448
  Male | 2754 | 2674 | 5428

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of SDB in Chronic HF Patients
Description: SDB= Sleep disordered breathing; HF= Heart failure
Time Frame: 1 night: Patients fulfilling the inclusion and exclusion criteria were examined for sleep-disordered breathing during 1 night in a sleep facility
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic HF With SDB
Number analyzed (Participants) | 6876
Participants | 3190

2. Secondary Outcome: Left Ventricular Ejection Fraction
Description: Amount of blood in the left ventricle at the end of Diastole that is being pumped into the System during systole
Time Frame: 1 night: Patients fulfilling the inclusion and exclusion criteria were examined for LVEF in a medical institution
Measure: Mean (Standard Deviation); unit: % ejection fraction
Arm/Group | Chronic HF Without SDB | Chronic HF With SDB
Number analyzed (Participants) | 3686 | 3190
% ejection fraction | 33.6 (8.0) | 32.8 (8.3)

3. Secondary Outcome: Age
Description: Age years
Time Frame: 1-time single assessment at baseline
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Chronic HF Without SDB | Chronic HF With SDB
Number analyzed (Participants) | 3686 | 3190
years | 65 (12) | 69 (11)

4. Secondary Outcome: Body Mass Index
Time Frame: 1-time single assessment at baseline
Measure: Mean (Standard Deviation); unit: kg/m˄2
Arm/Group | Chronic HF Without SDB | Chronic HF With SDB
Number analyzed (Participants) | 3686 | 3190
kg/m˄2 | 28.1 (5.0) | 28.9 (5.2)

5. Secondary Outcome: Male Gender
Time Frame: 1-time single assessment at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic HF Without SDB | Chronic HF With SDB
Number analyzed (Participants) | 3686 | 3190
Participants | 2754 | 2674

6. Secondary Outcome: NYHA Class ≥III
Description: New York Heart Association Class III: Marked Limitation of physical activity. Comfortable at rest, but less than ordinary physical activity results in undue breathlessness, fatigue or palpitations.
Time Frame: At baseline, the NYHA was determined in a medical institution or taken restrospectively from medical records
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic HF Without SDB | Chronic HF With SDB
Number analyzed (Participants) | 3686 | 3190
Participants | 2566 | 2341

7. Secondary Outcome: Ischemic Etiology
Description: Ischemic etiology describes a condition where a weakening or disease of the heart muscle is caused by reduced supply of blood (underlying cause might be the coronary artery). Secondary outcome ischemic etiology describes the cause of heart failure (HF) "ischemic" in HF patients without and with sleep-disordered breathing in percent of the respective study arm/group: e.g. x% of patients without SDB have HF with an ischemic etiology.
Time Frame: 1-time: At baseline the ischemic etiology was determined in the medical institution or taken retrospectively from the medical records.
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic HF Without SDB | Chronic HF With SDB
Number analyzed (Participants) | 3686 | 3190
Participants | 1961 | 1742

8. Secondary Outcome: Atrial Fibrillation
Time Frame: 1-time: At baseline atrial fibrillation (AF) was determined in the medical institution or AF history was taken retrospectively from the medical records
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic HF Without SDB | Chronic HF With SDB
Number analyzed (Participants) | 3686 | 3190
Participants | 863 | 1001

9. Secondary Outcome: Nocturnal Dyspnea
Time Frame: 1-time: At baseline history of nocturnal dyspnea taken retrospectively from the medical records
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic HF Without SDB | Chronic HF With SDB
Number analyzed (Participants) | 3686 | 3190
Participants | 672 | 800

10. Secondary Outcome: Nocturia ≥3 Times/Night
Time Frame: 1-time: At baseline nocturia was assessed 1 time (anamnesis)
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic HF Without SDB | Chronic HF With SDB
Number analyzed (Participants) | 3686 | 3190
Participants | 580 | 660

11. Secondary Outcome: Apnoea-Hypopnea-Index
Description: Number of Apnoeas (cessation of airflow for at least 10 seconds) and hypopneas (reduced airflow for at least 10 seconds) per hours of sleep
Time Frame: 1 night: Apnoea-Hypopnea Index (AHI) was assessed during one night under polysomnography (PSG) in a sleep facility
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | Chronic HF Without SDB | Chronic HF With SDB
Number analyzed (Participants) | 3686 | 3190
events/hour | 6 (4) | 31 (14)

12. Secondary Outcome: Oxygen Desaturation Index
Description: Number of times that arterial blood oxygen saturation Drops by ≥3% from the Basic value.
Time Frame: 1 time: Oxygen desaturation Index (ODI) was assessed during one night under polysomnography (PSG) in a sleep facility
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | Chronic HF Without SDB | Chronic HF With SDB
Number analyzed (Participants) | 3686 | 3190
events/hour | 8 (10) | 24 (15)

13. Secondary Outcome: Mean SpO2
Description: Saturation of oxygen
Time Frame: 1 night: oxygen saturation was assessed during one night under polysomnography (PSG) in a sleep facility
Measure: Mean (Standard Deviation); unit: %oxygen saturation
Arm/Group | Chronic HF Without SDB | Chronic HF With SDB
Number analyzed (Participants) | 3686 | 3190
%oxygen saturation | 93 (2) | 92 (3)

14. Secondary Outcome: Min SpO2
Description: Lowest Saturation with oxygen
Time Frame: 1 night: Minimum saturation with oxygen was assessed during one night under polysomnography (PSG) in a sleep facility
Measure: Mean (Standard Deviation); unit: % oxygen saturation
Arm/Group | Chronic HF Without SDB | Chronic HF With SDB
Number analyzed (Participants) | 3686 | 3190
% oxygen saturation | 83 (6) | 80 (6)

15. Secondary Outcome: Medication ACE Inhibitors and/ARBs
Description: ACE: Angiotensin converting Enzyme; ARB Angiotension receptor blocker
Time Frame: 1-time: At baseline medication was assessed 1 time (anamnesis)
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic HF Without SDB | Chronic HF With SDB
Number analyzed (Participants) | 3686 | 3190
Participants | 3269 | 2812

16. Secondary Outcome: Beta-blocker
Time Frame: 1-time: At baseline medication was assessed 1 time (anamnesis)
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic HF Without SDB | Chronic HF With SDB
Number analyzed (Participants) | 3686 | 3190
Participants | 3284 | 2824

17. Secondary Outcome: Diuretics
Time Frame: 1-time: At baseline medication was assessed 1 time (anamnesis)
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic HF Without SDB | Chronic HF With SDB
Number analyzed (Participants) | 3686 | 3190
Participants | 2805 | 2617

18. Secondary Outcome: Digitalis
Time Frame: 1-time: At baseline medication was assessed 1 time (anamnesis)
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic HF Without SDB | Chronic HF With SDB
Number analyzed (Participants) | 3686 | 3190
Participants | 717 | 599

19. Secondary Outcome: Aldosterone Antagonists
Time Frame: 1-time: At baseline medication was assessed 1 time (anamnesis)
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic HF Without SDB | Chronic HF With SDB
Number analyzed (Participants) | 3686 | 3190
Participants | 1808 | 1454

20. Secondary Outcome: Male Gender as Predictor for SDB in Chronic HF
Description: From the total number of participants, the number of male patients without and with SDB were counted and an odds Ratio for male sex as predictor for SDB in chronic heart failure
Time Frame: 1-time: At baseline physical status was assessed 1 time (anamnesis and medical records)
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Chronic HF Without SDB Male: patients with chronic heart failure and no sleep disordered breathing who are male
- Patients With Chronic Heart Failure and SDB Male: patients with chronic heart failure and sleep disorderd breathing who are male
Arm/Group | Patients With Chronic HF Without SDB Male | Patients With Chronic Heart Failure and SDB Male
Number analyzed (Participants) | 3686 | 3190
Participants | 2754 | 2674
Statistical Analysis 1: Comparison: Patients With Chronic HF Without SDB Male vs Patients With Chronic Heart Failure and SDB Male; Test type: Other; Odds Ratio (OR) = 1.90

21. Secondary Outcome: Atrial Fibrillation (AF) as a Predictor for SDB in Chronic HF
Description: From the total number of participants, the number of male patients without and with SDB were counted and an odds ratio calculated for AF as predictor for SDB in chronic heart failure
Time Frame: 1-time: At baseline physical status was assessed 1 time (anamnesis and medical records)
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Chronic HF Without SDB and AF: patients with chronic heart failure and no sleep disordered breathing who have atrial fibrillation (AF)
- Patients With Chronic Heart Failure and SDB and AF: patients with chronic heart failure and sleep disorderd breathing who have atrial fibrillation (AF)
Arm/Group | Patients With Chronic HF Without SDB and AF | Patients With Chronic Heart Failure and SDB and AF
Number analyzed (Participants) | 3686 | 3190
Participants | 863 | 1001
Statistical Analysis 1: Comparison: Patients With Chronic HF Without SDB and AF vs Patients With Chronic Heart Failure and SDB and AF; Test type: Other; Odds Ratio (OR) = 1.19

22. Secondary Outcome: Ischemic Etiology as Predictor for SDB in Chronic HF
Description: From the total number of participants, the number of male patients without and with SDB were counted and an odds ratio calculated for ischemic etiology as predictor for SDB in chronic heart failure
Time Frame: 1-time: At baseline physical status was assessed 1 time (anamnesis and medical records)
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Chronic HF Without SDB and Ischemic Etiology: patients with chronic heart failure and no sleep disordered breathing who have an ischemic etiology (reduced blood flow to the heart muscle) of HF
- Patients With Chronic Heart Failure and SDB and Ischemic Etiol: patients with chronic heart failure and sleep disorderd breathing who have an ischemic etiology (reduced blood flow to the heart muscle) of HF
Arm/Group | Patients With Chronic HF Without SDB and Ischemic Etiology | Patients With Chronic Heart Failure and SDB and Ischemic Etiol
Number analyzed (Participants) | 3686 | 3190
Participants | 1961 | 1742
Statistical Analysis 1: Comparison: Patients With Chronic HF Without SDB and Ischemic Etiology vs Patients With Chronic Heart Failure and SDB and Ischemic Etiol; Test type: Other; Odds Ratio (OR) = 0.92

23. Secondary Outcome: NYHA Class >= III as Predictor for SDB in Chronic HF
Description: From the total number of participants, the number of male patients without and with SDB were counted and an odds ratio calculated for NYHA (New York Heart Association - class I not impaired, class II slighly impaired, class III severly impaired, class IV = unable to perform normal tasks) class≥III as predictor for SDB in chronic heart failure
Time Frame: 1-time: At baseline physical status was assessed 1 time (anamnesis and medical records)
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Chronic HF Without SDB and NYHA>III: patients with chronic heart failure and no sleep disordered breathing who are classified as NYHA >=III
- Patients With Chronic Heart Failure and SDB and NYHA >III: patients with chronic heart failure and sleep disorderd breathing who are classified as NYHA >=III
Arm/Group | Patients With Chronic HF Without SDB and NYHA>III | Patients With Chronic Heart Failure and SDB and NYHA >III
Number analyzed (Participants) | 3686 | 3190
Participants | 2566 | 2341
Statistical Analysis 1: Comparison: Patients With Chronic HF Without SDB and NYHA>III vs Patients With Chronic Heart Failure and SDB and NYHA >III; Test type: Other; Odds Ratio (OR) = 1.12

ADVERSE EVENTS:
Description: Non-serious adverse events were not collected in this observational study. Usual side-effects of therapy in clinical routine are well described. Serious adverse events (SAE) were recorded, but in this observational study only those in connection to the device: Unexpected serious device defects (USADE). No device effects were recorded during the course of this study.
Arm/Group | Chronic HF Without SDB | Chronic HF With SDB
Serious Adverse Events (participants affected / at risk) | 0/3686 | 0/3190
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No